CLINICAL TRIAL: NCT02095925
Title: Microparticle's Procoagulant Activity to Identify Patients With Cancer and a High Risk for Venous Thrombosis
Brief Title: Cohort Study to Identify Cancer Patients at High Risk of Venous Thromboembolism
Acronym: MICA
Status: Completed | Type: Observational
Sponsor: Harry R. Buller (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amsterdam UMC, location VUmc (Other); University Medical Center Groningen (Other); Slotervaart Hospital (Other); Hôpital Louis Mourier (Other); Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other); Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Sponsor-Investigator, Harry R. Buller, Harry R Büller, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: MICA
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cancer; Deep Venous Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Neoplasms; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — citrated plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cancer patients: Patients with stage III or IV esophageal carcinoma, gastric carcinoma, intestinal carcinoma, pancreatic carcinoma, ovarian cancer, breast carcinoma, prostate cancer, urothelial cell carcinoma or lung carcinoma (small cell or non-small cell) who have started chemotherapy no more than 3 months ago

SUMMARY:
Cancer patients are at increased risk of deep venous thrombosis and pulmonary embolism, collectively termed venous thromboembolism (VTE). Risk assessment scores for VTE in cancer patients have been previously developed by the groups of Khorana and Vienna CATS. However, routine thromboprophylaxis for ambulatory cancer patients based on these scores is currently not recommended. In the investigators prospective, observational cohort study, the investigators aim to identify cancer patients at high risk for VTE based on clinical characteristics, coagulation biomarkers and the coagulant activity of tissue factor bearing microparticles.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV esophageal carcinoma, gastric carcinoma, intestinal carcinoma, pancreatic carcinoma, ovarian cancer, breast carcinoma, prostate cancer, urothelial cell carcinoma or lung carcinoma (small cell or non-small cell) who have started chemotherapy no more than 3 months ago
* Chemotherapy started no more than 3 months ago or within 7 days after enrollment
* Aged 18 years or older
* Written informed consent

Exclusion Criteria:

* Use of anticoagulants (heparin, vitamin K antagonists or direct oral anticoagulants)
* Adjuvant chemotherapy (i.e. after surgery with curative intent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III or IV esophageal carcinoma, gastric carcinoma, intestinal carcinoma, pancreatic carcinoma, ovarian cancer, breast carcinoma, prostate cancer, urothelial cell carcinoma or lung carcinoma (small cell or non-small cell) who have started chemotherapy no more than 3 months ago
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2008-07; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
venous thromboembolism | 6 months after enrollment
  Objectively confirmed asymptomatic or symptomatic deep venous thrombosis or pulmonary embolism

SECONDARY OUTCOMES:
all-cause mortality | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Harry R Buller, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (7):
- Hopital Louis Mourier, Colombes, Île-de-France Region, France
- Hospital D'Annunziata, Chieti, Italy
- Instituto Nacional de Cancerología, Mexico City, Mexico
- Netherlands (4):
  - Slotervaart hospital, Amsterdam, North Holland
  - VU medical center, Amsterdam, North Holland
  - Academic Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen, Provincie Groningen

REFERENCES:
- [Derived] van Es N, Di Nisio M, Cesarman G, Kleinjan A, Otten HM, Mahe I, Wilts IT, Twint DC, Porreca E, Arrieta O, Stepanian A, Smit K, De Tursi M, Bleker SM, Bossuyt PM, Nieuwland R, Kamphuisen PW, Buller HR. Comparison of risk prediction scores for venous thromboembolism in cancer patients: a prospective cohort study. Haematologica. 2017 Sep;102(9):1494-1501. doi: 10.3324/haematol.2017.169060. Epub 2017 May 26. PMID 28550192